CLINICAL TRIAL: NCT05853822
Title: FirmTech User Research Trial
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Collaborators: FirmTech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Firmtech_RMANJ_01
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Erectile Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: FirmTech Tech Ring — Participants will utilize the FirmTech Tech Ring at least twice during a two-week time period and complete a survey
Other: Giddy Penile Constriction Ring — Participants will utilize the Giddy Penile Constriction at least twice during a two-week time period and complete a survey

SUMMARY:
The objective of this study is to see whether a home-use penile constriction device, Firmtech Tech Ring, can be determined to be superior to the Giddy device through evaluation of Leikert scale scores to assess ease of use and participant comfort and satisfaction with erectile quality with these devices. The primary outcome will be the satisfaction with use of the device as assessed through the Leikert scores. The other outcomes will be secondary.

ELIGIBILITY:
Inclusion Criteria:

* All English-speaking participants > 18 years old recruited through social media.
* Physically and emotionally capable of engaging in sexual activity with at least one attempt per week of masturbation or sexual intercourse

Exclusion Criteria:

* Men who cannot understand English.
* Men with a prior or current penile implant.
* Transgender or non-binary individuals
* Men diagnosed with a hidden or buried penis.
* Investigator's impression of expected poor participant compliance or anatomic inadequacy (penile size/girth)
* Any psychiatric disorder, which, in the opinion of the investigator, would prohibit participation.
* Coagulopathy or other blood disorder which the investigator determines would affect the participant's participation in the trial.
* Any tumor in the pelvic or penile region within the last 3 years
* Men with an active caregiver who are unable to live independently.
* Men who the provider is concerned would be at high risk for non-healing wounds of the penis.
* Participants with sensory disorders like sensory processing disorder, sensory integration dysfunction disorder, neuropathies, etc.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample from social media recruitment
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Device satisfaction via Leikert scores | 2 weeks after receiving device
  A survey will be completed for each device after utilization

CONTACTS AND LOCATIONS:
Locations (1):
- IVI RMA New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rendon DO, Saffati G, Whitehead C, Zuckerman C, Hom A, Daily R, Khera M, Cheng PJ. Penile constriction devices: a randomized survey study to compare preferences between two medical-grade devices. J Sex Med. 2025 Jan 3;22(1):43-50. doi: 10.1093/jsxmed/qdae151. PMID 39545359